CLINICAL TRIAL: NCT00914056
Title: Is Continuous Lactulose Therapy Necessary for Patients With Hepatic Encephalopathy? A Prospective Study of Controlled Lactulose Withdrawal
Brief Title: A Study of Controlled Lactulose Withdrawal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jasmohan Bajaj, Associate Professor of Medicine, Hunter Holmes Mcguire Veteran Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Bajaj 006
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Lactulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lactulose withdrawal (Experimental): Patients who were started on lactulose as a result of a precipitated HE episode underwent analysis while they were on lactulose; after this they underwent a controlled lactulose withdrawal with 3 visits post-withdrawal at 2 days, 14 days and 30 days after lactulose withdrawal
  Interventions: Drug: lactulose

INTERVENTIONS:
Drug: lactulose — withdrawal of lactulose

SUMMARY:
After resolution of the initial episode of hepatic encephalopathy (HE), lactulose is routinely continued indefinitely as maintenance therapy. Although widely used for this indication, lactulose has never been shown in randomized, controlled trials to be effective for preventing exacerbations of HE. Indeed, lactulose was found to be ineffective at preventing HE when administered prophylactically to patients undergoing portosystemic shunt insertion. While some patients may be lactulose dependent following an initial episode of HE, it is likely that most could have their lactulose discontinued with no adverse consequences.

This goal is worth pursuing because lactulose is not innocuous. It has an unpleasant taste, and it routinely produces gastrointestinal symptoms, including bloating, gas and diarrhea. In high doses it can cause incontinence, dehydration and electrolyte derangements. Patients universally dislike taking lactulose and often are noncompliant with treatment. A recent trial showed that patients on lactulose had a substantial risk of hospital admissions due to lactulose-related complications and treatment non-compliance.

DETAILED DESCRIPTION:
In this pilot study we propose to perform controlled lactulose withdrawal in selected patients with HE whose initial presentation follows a clearly defined, reversible precipitating event or those with stable, chronic HE. We hypothesize that a majority of these patients can be withdrawn from daily lactulose therapy without deterioration of cognitive function, and that lactulose withdrawal will improve symptoms and quality of life for these individuals. We propose to carry out a comprehensive battery of clinical, laboratory, microbiological and psychometric evaluations before and after lactulose withdrawal. We will closely follow changes in cognitive function and re-institute lactulose therapy at the first sign of clinical deterioration. Through multivariate analysis we propose to develop a model to discriminate between treatment dependent and treatment independent patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hepatic cirrhosis based on biopsy, clinical and/or radiological findings.
* Stable HE (chronic): On daily lactulose for more than 6 months without hospitalization for HE within 3 months of enrollment.
* Treated with lactulose on a daily basis, with restoration of mental status to baseline.
* Lives with an adult individual who is willing to serve as a full-time caregiver.
* Able and willing to give informed consent.

Exclusion Criteria:

* Use of antibiotics, including rifaximin.
* Patient without an adult caregiver.
* Pre-existing focal neurological deficits, seizures or other indication of structural neurological disorder.
* Actively abusing illicit drugs or alcohol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-09; Primary Completion 2009-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Psychometric function and relapse into clinical HE | 30 days

SECONDARY OUTCOMES:
MR Spectroscopy | 30 days
Pro-inflammatory cytokines | 30 days
Stool bacterial DNA analysis | 30 days
Urine and blood for metabolomics | 30 days
Quality of life | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

REFERENCES:
- [Result] Bajaj JS, Gillevet PM, Patel NR, Ahluwalia V, Ridlon JM, Kettenmann B, Schubert CM, Sikaroodi M, Heuman DM, Crossey MM, Bell DE, Hylemon PB, Fatouros PP, Taylor-Robinson SD. A longitudinal systems biology analysis of lactulose withdrawal in hepatic encephalopathy. Metab Brain Dis. 2012 Jun;27(2):205-15. doi: 10.1007/s11011-012-9303-0. Epub 2012 Apr 12. PMID 22527995
- [Result] Bajaj JS, Ridlon JM, Hylemon PB, Thacker LR, Heuman DM, Smith S, Sikaroodi M, Gillevet PM. Linkage of gut microbiome with cognition in hepatic encephalopathy. Am J Physiol Gastrointest Liver Physiol. 2012 Jan 1;302(1):G168-75. doi: 10.1152/ajpgi.00190.2011. Epub 2011 Sep 22. PMID 21940902